CLINICAL TRIAL: NCT02158767
Title: Access Protocol. Infusion of CD34+ Enriched, T Cell Depleted Hematopoietic Stem Cell Grafts.
Status: No longer available | Type: Expanded Access
Sponsor: Leland Metheny (Other)
Responsible Party: Sponsor-Investigator, Leland Metheny, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Other Study IDs: CASE16Z13
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Hematologic Neoplasms

INTERVENTIONS:
Biological: Allogenic T cell-depleted hematopoietic stem cell transplantation — Undergo CD34+ enriched T-cell depleted allogeneic peripheral blood stem cell transplant. T-cells will be removed using the experimental CliniMACS(r) Reagent System used in vitro to select and enrich CD34+ cells

SUMMARY:
This clinical trial studies the use of a second infusion of donor hematopoietic cells that have had removal of T cells for the treatment of engraftment failure after a first hematopoietic stem cell transplant.

Hematopoietic cell transplants from donors can be complicated by complete or incomplete failure of recovery of blood counts. This results in frequent needs for transfusions and other methods to maintain blood counts at acceptable levels. One way of improving the blood counts in the recipient is to give a "booster" dose of cells from the donor, but this is associated with increased risk of an immune reaction from the donor cells against the recipient cells. To decrease this risk, it is possible to decrease the amount of T cells, responsible for this type of immune reaction. These cells are removed by a special handling of the graft, which allows to remove the cells directly or indirectly (by selecting other cells to "stay" in the graft").

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide patients with suboptimal engraftment after allogeneic stem cell transplantation access to donor - derived, cluster of differentiation (CD34)+ enriched or T-cell depleted peripheral blood stem cells isolated by the CliniMACS System.

OUTLINE:

Patients undergo CD34+ enriched or T-cell depleted peripheral blood stem cell infusion (PBSCT) over 1-3 hours.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a prior hematopoietic progenitor cell transplantation, including matched sibling and unrelated donor transplants, mismatched sibling and unrelated donor transplants and haploidentical transplants from related donors
* Patients with a presence of secondary engraftment failure defined as decrease in donor chimerism by ≥ 50% (i.e. 40% to 20%) in two measurements done at least 30 days apart
* OR a presence of incomplete graft function manifested by presence of persistent or new cytopenias 60 or more days after transplantation:

  * Anemia; hemoglobin less than 8g/dL, or red blood cell transfusion requirements over the preceding 4 weeks
  * Neutropenia, with absolute neutrophil count less than 1,000 neutrophils per microliter or requirement of growth factor support over the preceding 4 weeks
  * Thrombocytopenia, with platelet counts below 20,000 platelets per microliter or platelet transfusion requirements over the preceding 4 weeks

Exclusion Criteria:

* Patients for whom hematopoietic progenitor cells from the original donor are not available
* Presence of reversible causes of engraftment failure or incomplete graft function, including

  * Active viral infection
  * Medications
  * Acute or chronic graft versus host disease (GVHD) that is not controlled to less or equal than stage II with immunosuppressants

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States